CLINICAL TRIAL: NCT04156087
Title: Progression-free Survival After Minimally Invasive Surgical Microwave Ablation Plus Durvalumab (MEDI4736) and Tremelimumab for Unresectable Non-metastatic Locally Advanced Pancreatic Cancer: MIMIPAC Trial
Brief Title: Progression-free Survival After MWA Plus Durvalumab and Tremelimumab for Unresectable Locally Advanced Pancreatic Cancer
Acronym: MIMIPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baki Topal (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Baki Topal, Professor, Doctor, University Hospital, Gasthuisberg
Organization: University Hospital, Gasthuisberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZ S61508; 2018-002852-34 (EudraCT Number)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer Non-resectable
MeSH Terms: interventions — durvalumab; tremelimumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MIMIPAC (Experimental): Intervention: MIS-MWA plus immunotherapy using the combination of durvalumab with tremelimumab
  Interventions: Drug: Durvalumab 50 MG/ML; Drug: Tremelimumab; Drug: Gemcitabine; Procedure: Minimally Invasive Surgical Microwave Ablation (MIS-MWA)

INTERVENTIONS:
Drug: Durvalumab 50 MG/ML — Combination of Durvalumab (fixed dose of 1500 mg) and Tremelimumab (fixed dose of 75 mg) will be given 2 weeks before surgery.
  Minimally invasive surgical microwave ablation (MIS-MWA) of the pancreatic tumor will be performed two weeks after the first dose of Durvalumab and Tremelimumab After 4 doses of Durvalumab and Tremelimumab, only Durvalumab 1500mg is provided q4w until disease progression.
  Systemic gemcitabine will be started 6 weeks after MIS-MWA. Gemcitabine will be given at a dose of 1000 mg /m² body surface, once a week for 3 weeks, followed with a week of rest.
  Other Names: MEDI4736; IMFINZI
Drug: Tremelimumab — Combination of Durvalumab (fixed dose of 1500 mg) and Tremelimumab (fixed dose of 75 mg) will be given 2 weeks before surgery.
  Minimally invasive surgical microwave ablation (MIS-MWA) of the pancreatic tumor will be performed two weeks after the first dose of Durvalumab and Tremelimumab After 4 doses of Durvalumab and Tremelimumab, only Durvalumab 1500mg is provided q4w until disease progression.
  Systemic gemcitabine will be started 6 weeks after MIS-MWA. Gemcitabine will be given at a dose of 1000 mg /m² body surface, once a week for 3 weeks, followed with a week of rest.
Drug: Gemcitabine — Combination of Durvalumab (fixed dose of 1500 mg) and Tremelimumab (fixed dose of 75 mg) will be given 2 weeks before surgery.
  Minimally invasive surgical microwave ablation (MIS-MWA) of the pancreatic tumor will be performed two weeks after the first dose of Durvalumab and Tremelimumab After 4 doses of Durvalumab and Tremelimumab, only Durvalumab 1500mg is provided q4w until disease progression.
  Systemic gemcitabine will be started 6 weeks after MIS-MWA. Gemcitabine will be given at a dose of 1000 mg /m² body surface, once a week for 3 weeks, followed with a week of rest.
  Other Names: Gemzar
Procedure: Minimally Invasive Surgical Microwave Ablation (MIS-MWA) — Minimally invasive surgical microwave ablation (MIS-MWA) of the pancreatic tumor will be performed two weeks after the first dose of Durvalumab and Tremelimumab

SUMMARY:
This phase-2 monocenter non-randomized prospective clinical trial evaluates the effectiveness of minimally invasive microwave ablation plus immunotherapy for unresectable non-metastatic locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Research Hypothesis Does MIS-MWA combined with durvalumab (MEDI4736) plus tremelimumab and gemcitabine prolong progression-free survival in patients with unresectable non-metastatic adenocarcinoma of the pancreas?

Investigational Product(s) and Reference Therapy:

Combination of Durvalumab (fixed dose of 1500 mg) and Tremelimumab (fixed dose of 75 mg) will be given 2 weeks before surgery.

Minimally invasive surgical microwave ablation (MIS-MWA) of the pancreatic tumor will be performed two weeks after the first dose of Durvalumab and Tremelimumab After 4 doses of Durvalumab and Tremelimumab, only Durvalumab 1500mg is provided q4w until disease progression.

Systemic gemcitabine will be started 6 weeks after MIS-MWA. Gemcitabine will be given at a dose of 1000 mg /m² body surface, once a week for 3 weeks, followed with a week of rest.

Objectives:

Primary Objectives:

Progression-free survival (PFS)

Secondary Objectives:

* Safety: clinical and hematological toxicity (NCI CTCAE v. 5.0) of chemotherapy and immunotherapy
* Safety: number and type of postoperative complications of the MIS-MWA procedure
* Length of hospital stay

Tertiary Objectives Overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable non-metastatic Locally Advanced Pancreatic Cancer (LAPC) defined according to NCCN guidelines Version 2.2017
* Histologically proven adenocarcinoma of the pancreas located in the head, body or tail
* LAPC tumor greatest diameter maximum 5 cm
* Male or female, age 18 years and older, ECOG PS 0-1
* Life expectancy of at least 12 weeks
* Only patients who did not receive chemotherapy for their PC are allowed
* Patients without distant organ metastases on conventional diagnostic imaging
* Pre-operative biliary drainage for obstructive jaundice is allowed, but the type of biliary stent is standardized in all jaundiced patients
* Patients fit for MIS-MWA
* Able to receive Durvalumab and Tremelimumab.
* Patients with good liver and renal function and with good hematology
* Effective contraception for both male and female patients if applicable. Women of childbearing potential must have negative blood pregnancy test at screening visit.
* Written informed consent (+ optional for TR) must be given according to ICH/GCP and national/European regulations

Exclusion Criteria:

* Pregnancy
* Metastatic PC on conventional diagnostic imaging or staging laparoscopy
* LAPC tumor greatest diameter is larger than 5 cm
* Borderline or resectable PC defined according to the NCCN guidelines version 2.2017
* Systemic chemo(radio)therapy is not allowed before MIS-MWA
* Major surgical procedure within 28 days prior to the first dose of investigational products
* Classic contraindications for PDL and CTLA antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  The study is exploratory and cannot be statistically powered for comparisons. Median progression-free survival (PFS) time is chosen as the clinically meaningful outcome. Survival estimates will be calculated using the Kaplan-Meier method. For information, the reference PFS time in patients with non-metastatic LAPC treated with gemcitabine monotherapy is about 6 months. Results will be presented descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No